CLINICAL TRIAL: NCT01660555
Title: The Real Distribution of Microbiota Along the Colonic Mucosa Using a Novel Device Capable of Taking 'Protected' Biopsies
Brief Title: The Real Distribution of Microbiota Along the Colon Using a Novel Device Along the Colon Using a Novel Device
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, C.Y. Ponsioen, MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: METC 2011_026#C201136
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Patients Scheduled for Colonoscopy
Keywords: Microbiota; HITChip; biopsies; colon; protected biopsies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — mucosal biopsies will be screened for diversity by Denaturing Gradient Gel Electrophoresis of 16S rRNA genes and subsequently analysed with the HITChip.
  (-> DNA from microbiota instead of human DNA will be analysed)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patiënts scheduled for colonoscopy: Ill prepared colon during index colonoscopy or sigmoidoscopy: Boston scale <3

SUMMARY:
The human microbiota forms a highly complex ecosystem with its host, consisting of hundreds of different species of microorganisms, the majority of which have not yet been cultured. With the recent advent of small subunit rRNA (SSU rRNA) gene sequencing technology, it is estimated that the number of specific gastrointestinal tract phylotypes is more than 1800. Sampling techniques might constitute a major confounder in the read-out of highly sensitive techniques such as SSU-DNA analysis.

It is not properly established whether there is a difference in distribution of luminal bacteria or mucosa adherent bacteria proximal or distal in the colon. In addition, 'bowel lavage' before endoscopy might result in a disturbance of the microbiota in the bowel. For this proof of concept study a novel device capable of taking 'protected' biopsies has been designed.

We hypothesize that the distribution of mucosal and luminal microbiota changes from proximal to distal in the colon, and by taking 'protected biopsies' there will be the opportunity to show the real distribution of microbiota according to the localisation in the colon.

Furthermore, we hypothesize that microbial diversity will differ after bowel lavage.

DETAILED DESCRIPTION:
We hypothesize that the distribution of mucosal and luminal microbiota changes from proximal to distal in the colon, and by taking 'protected biopsies' there will be the opportunity to show the real distribution of microbiota according to the localisation in the colon.

ELIGIBILITY:
* Inclusion Criteria:

  * Ill prepared colon during index colonoscopy or sigmoidoscopy: Boston scale <3
* Sufficient indication to perform colonoscopy again

Exclusion Criteria:

* Inability to give informed consent
* Life expectancy < 12 months
* Use of combination of two platelet aggregation inhibitors
* Mandatory use of anti-coagulatory medication
* Known history of hemostatic disorder
* Use of systemic antibiotics in preceding 6 weeks
* Use of probiotic or prebiotic treatment in preceding 6 weeks
* Positive stool cultures for common enteric pathogens (Salmonella, Shigella, Yersinia, Campylobacter, enteropathogenic e coli)
* History of surgery:

  * Resection of any part of the colon or Ileocoecal resection
  * Presence of an ileo- or colostoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatients scheduled for colonoscopy for diagnostical purposes who are not known with infectious enterocolitis.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Intra-individual differences in phylogenetic fingerprinting and phylotype quantification from mucosal and faecal biopsy samples located at the colon ascendens and the sigmoid both in an 'ill prepared' as well as in a 'well-prepared' situation | at baseline colonoscopy, and if the colonoscopy will be repeated
  'ill-prepared' patients will be included, biopsies will be taken at baseline colonoscopy.
  patients will be re-scheduled, and better prepared with laxatives for the 2nd colonoscopy: biospies will be taken again.

SECONDARY OUTCOMES:
Intra-individual differences in phylogenetic fingerprinting and phylotype quantification from mucosal and faecal biopsy samples located at the colon ascendens and sigmoid using 'protected' biopsy material versus 'un-protected' material. | at baseline colonoscopy, and if the colonoscopy will be repeated
  'ill-prepared' patients will be included, biopsies will be taken at baseline colonoscopy.
  patients will be re-scheduled, and better prepared with laxatives for the 2nd colonoscopy: biospies will be taken again.

CONTACTS AND LOCATIONS:
Overall Officials: CY Ponsioen, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (2):
- Netherlands (2):
  - Academic medical Center, Amsterdam
  - Academic_Medical_Center, Amsterdam